CLINICAL TRIAL: NCT01806922
Title: Yoga Exercise for Improving Balance in Patients With Subacute &Ｃhronic Stroke : A Pilot Study
Brief Title: Yoga Exercise for Improving Balance in Patients With Subacute &Ｃhronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201210006RIB
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Depression; Stroke
Keywords: Yoga; Stroke; Standing balance; Depression
MeSH Terms: conditions — Depression; Stroke | interventions — Yoga

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga training, Tradiational physiotherapy (Experimental): Experimental Group(20 people) receive tradiational physiotherapy(4 times in a week, every time 1 hour), and 8-weeks yoga training(2 time in a week, every time 1 hour)
  Interventions: Behavioral: Yoga
- Tradiational physiotherapy (No Intervention): Control Group(20 people)only receive tradiational rehabiliation( 4 times in a week, every time 1 hour ) for 8 weeks.

INTERVENTIONS:
Behavioral: Yoga
  Arms: Yoga training, Tradiational physiotherapy

SUMMARY:
Hypothesis: This study investigated the hypothesis that subacute and chronic stroke patients who received a combination of yoga and traditional physiotherapy were getting more improvement in standing balance than traditional physiotherapy. And we also hypothesis yoga can improve post-stroke depression symtom.

ELIGIBILITY:
Inclusion Criteria:

1. The time of stroke onset is more than 91 days.
2. Able to stand for more than 1 minutes.
3. Between the ages of 30 and 80.

Exclusion Criteria:

1. Now receive others palliative therapy.
2. Significant psychotic disease.
3. Obvious language disorder.
4. Medical contraindication(clincans evaluate cannot included).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Berg Balance Scale | within 7 days after finish yoga therapy course

SECONDARY OUTCOMES:
Taiwanese Depression Questionnaire | within 7 days after finish yoga therapy course

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ting Lai, Principal Investigator — National Taiwan University Hospital Hsin-Chu Branch
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Taoyuan District, Taiwan

REFERENCES:
- [Background] 1.Tyson SF, Hanley M, Chillala J, Selley A, Tallis RC. Balance disability after stroke. Phys Ther. 2006;86:30. 2.Jorgensen L, Engstad T, Jacobsen BK. Higher incidence of falls in long-term stroke survivors than in population controls: Depressive symptoms predict falls after stroke. Stroke. 2002;33:542-547 3.Balance retraining after stroke using force platform biofeedback. Phys Ther. 1997 ; 77;553-58. 4.A yoga-based exercise program for people with chronic poststroke hemiparesis. Bastille JV, Gill-Body KM. Phys Ther. 2004 Jan;84(1):33-48. 5.Poststroke balance improves with yoga: a pilot study.Schmid AA, Van Puymbroeck M, Altenburger PA, Schalk NL, Dierks TA, Miller KK, Damush TM, Bravata DM, Williams LS. Stroke. 2012 Sep;43(9):2402-7. Epub 2012 Jul 26. 6.Chan W, Immink MA, Hillier S. Yoga and exercise for symptoms of depression and anxiety in people with poststroke disability: a randomized, controlled pilot trial. Altern Ther Health Med. 2012 May-Jun;18(3):34-43.